CLINICAL TRIAL: NCT02608736
Title: Phase 0 Clinical Trial With Valproic Acid as a Chemopreventive Agent in Patients With Head and Neck Squamous Cell Carcinoma Previously Treated
Brief Title: Chemoprevention of Head and Neck Squamous Cell Carcinoma (HNSCC) With Valproic Acid
Acronym: GAMA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BarretosCH - Head and Neck
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2016-09

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: head and neck squamous cell carcinoma; histone deacetylases; valproic acid; acetylation; chemoprevention; DNA methyltransferase; methylation
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valproic Acid (Experimental): Valproic acid will be orally administered in a total dose of 1500mg per day (500mg, every 8 hours), for three months.
  Interventions: Drug: Valproic Acid
- Placebo (Placebo Comparator): Placebo will be orally administered in a total dose of three capsules per day (every 8 hours), for three months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valproic Acid — Half of the participants will receive valproic acid orally for three months. Saliva and blood will be sampled in the study entry. The participants will be followed with blood tests every month for three cycles. After the third cycle, saliva and blood will be sampled once more. Finally, histone acetylation and DNMT expression will be studied comparing the samples collected in different timelines and comparing them to saliva collected in placebo arm.
  Other Names: Divalproex; Depakene; Depacon; Depakote
  Arms: Valproic Acid
Drug: Placebo — The other half of the participants will receive placebo for three months. Saliva and blood will be sampled in the study entry. The participants will be followed with blood tests every month for three cycles. After the third cycle, saliva and blood will be sampled once more. Finally, histone acetylation and DNMT expression will be studied comparing the samples collected in different timelines and comparing them to saliva collected in valproic acid arm.
  Other Names: Inert, not active
  Arms: Placebo

SUMMARY:
This study evaluates the addition of valproic acid as a chemopreventive drug in head and neck squamous cell carcinoma (HNSCC) patients that do not have signs of recurrence or residual disease. The participants will be randomized 1:1 (valproic acid : placebo). The primary outcome is to document histone acetylation and DNA methyltransferase expression (DNMT) in saliva collected from participants when comparing valproic acid arm with placebo arm.

DETAILED DESCRIPTION:
Chemoprevention is an attractive strategy to reduce the incidence of squamous cell carcinoma of the head and neck, although past trials have not demonstrated its feasibility.

Valproic acid (VA) is a modifier of epigenetic events as it is an histone deacetylase inhibitor and causes DNMT degradation. The histone deacetylase inhibitors (e.g. VA) encompasses a new class of anti-tumor drugs, that can affect multiple pathways related to tumor initiation and progression due to histone and non-histone protein acetylation and DNMT degradation. VA promote histone acetylation when orally administered with a dose of 20-40 mg/kg, per day or 1000/1500 mg, per day.

Initially the authors will study saliva from participants documenting if there is saliva histone acetylation and if a difference in DNMT expression in saliva exists when comparing valproic acid arm to placebo arm (biological validation) after giving placebo or valproic acid for three months.

This will be the initial step of a bigger project. If authors prove that there will be a difference in histone acetylation and/or DNMT expression between groups they will launch a randomized, double blind, placebo control clinical trial (phase 3 clinical trial), to evaluate VA action as a chemopreventive agent in HNSCC patients who usually carries a high chance to develop recurrence (stages III/IV) or second primary malignancies (stages I/II/III/IV).

ELIGIBILITY:
Inclusion Criteria:

* Patients that signed the formal consent;
* Previous history of head and neck squamous cell carcinoma with no more than three years of follow-up;
* History of squamous cell carcinoma in the following sub-sites: oral cavity, oropharynx, larynx and hypopharynx;
* Absence of active malignant disease (HNSCC) with at least three months of follow-up (without signs of residual disease, recurrence or second primary invasive tumors);
* Normal liver, hematologic and renal function.
* Eastern Cooperative Oncology Group (ECOG) Performance Status: 0, 1 or 2;
* Smoking history (current smokers or former smokers). Former users were defined as patients who had quit smoking at least one year prior to diagnosis and smoked more than 100 cigarettes in their lifetime.

Exclusion Criteria:

* Any active malignancy;
* History of invasive malignancies (other than HNSCC) diagnosed within the last 2 years (controlled non-melanoma skin cancer are an exception);
* History of hepatitis B, hepatitis C, HIV, chronic liver disease or chronic pancreatic disease;
* Any comorbid medical or psychiatric disorder that it is not well controlled;
* Patients under immunosuppression or under systemic corticosteroid therapy to treat any active autoimmune disease;
* Patients that still have documented toxicities greater than grade 1 (CTCEA NCI v4.0) due to the previously treated HNSCC;
* Patients that are pregnant or breast-feeding;
* Patients that are in routine use of the following medications due to drug interaction: phenytoin, carbamazepine, barbiturates, chlorpromazine, diazepam, clonazepam, lamotrigine, primidone, amitriptyline, nortriptyline, ethosuximide, warfarin, tolbutamide or topiramate;
* Any medical condition or mental disorder that can potentially increase their risk during the trial (e.g. epilepsy, active infection, schizophrenia);
* Patients that are already under valproic acid use due to neurological or psychiatric disorders;
* Patients that are allergic/intolerant to valproic acid;
* Patients with alcoholism history within the past year or that was under alcoholism treatment in the same period;
* Institutionalized patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Changes in protein or histone acetylation | Three months after study enrollment
  Saliva samples will be collected in baseline and three months after study enrolment. Histone acetylation will be quantified (through ELISA method) and compared in the same arm (if there will be a change in histone acetylation when looking at these different timelines) and between arms (if one group will have or will not have more histone acetylation than the other).

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Day 1 of each new cycle up to 3 months (3 months of treatment and 3 months of follow-up), in other words, from day 1 of the first cycle until the date of first documented emergent adverse event, assessed up to 6 months
  Evaluation of incidence of treatment-induced adverse events at the beginning of each new cycle (day 1, every 30 days, for a total of six months) using Common Toxicity Criteria for Adverse Effects (CTCAE v.4.0).
Change in DNA methyltransferases expression. (DNMT) | Three months after study enrollment
  Saliva samples will be collected in baseline and three months after study enrolment. DNA methyltransferases expression (through microarray method) will be compared in the same arm (if there will be a change in DNMT expression when looking at these different timelines) and between arms (if one group will have or will not have a different DNMT expression when compared to the other).

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Gama, MD, PHD, Principal Investigator — Barretos Cancer Hospital; André Lopes Carvalho, MD, PHD, Study Director — Barretos Cancer Hospital; Luciano de Souza Viana, MD, PHD, Study Chair — Barretos Cancer Hospital
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
As soon as we have results they will be shared.

REFERENCES:
- [Background] Brodie SA, Li G, El-Kommos A, Kang H, Ramalingam SS, Behera M, Gandhi K, Kowalski J, Sica GL, Khuri FR, Vertino PM, Brandes JC. Class I HDACs are mediators of smoke carcinogen-induced stabilization of DNMT1 and serve as promising targets for chemoprevention of lung cancer. Cancer Prev Res (Phila). 2014 Mar;7(3):351-61. doi: 10.1158/1940-6207.CAPR-13-0254. Epub 2014 Jan 17. PMID 24441677
- [Background] Gottlicher M, Minucci S, Zhu P, Kramer OH, Schimpf A, Giavara S, Sleeman JP, Lo Coco F, Nervi C, Pelicci PG, Heinzel T. Valproic acid defines a novel class of HDAC inhibitors inducing differentiation of transformed cells. EMBO J. 2001 Dec 17;20(24):6969-78. doi: 10.1093/emboj/20.24.6969. PMID 11742974
- [Background] Gan CP, Hamid S, Hor SY, Zain RB, Ismail SM, Wan Mustafa WM, Teo SH, Saunders N, Cheong SC. Valproic acid: growth inhibition of head and neck cancer by induction of terminal differentiation and senescence. Head Neck. 2012 Mar;34(3):344-53. doi: 10.1002/hed.21734. Epub 2011 Mar 24. PMID 21438066
- [Background] Chavez-Blanco A, Segura-Pacheco B, Perez-Cardenas E, Taja-Chayeb L, Cetina L, Candelaria M, Cantu D, Gonzalez-Fierro A, Garcia-Lopez P, Zambrano P, Perez-Plasencia C, Cabrera G, Trejo-Becerril C, Angeles E, Duenas-Gonzalez A. Histone acetylation and histone deacetylase activity of magnesium valproate in tumor and peripheral blood of patients with cervical cancer. A phase I study. Mol Cancer. 2005 Jul 7;4(1):22. doi: 10.1186/1476-4598-4-22. PMID 16001982
- [Background] Kang H, Gillespie TW, Goodman M, Brodie SA, Brandes M, Ribeiro M, Ramalingam SS, Shin DM, Khuri FR, Brandes JC. Long-term use of valproic acid in US veterans is associated with a reduced risk of smoking-related cases of head and neck cancer. Cancer. 2014 May 1;120(9):1394-400. doi: 10.1002/cncr.28479. Epub 2014 Mar 24. PMID 24664792
- [Background] Kuendgen A, Knipp S, Fox F, Strupp C, Hildebrandt B, Steidl C, Germing U, Haas R, Gattermann N. Results of a phase 2 study of valproic acid alone or in combination with all-trans retinoic acid in 75 patients with myelodysplastic syndrome and relapsed or refractory acute myeloid leukemia. Ann Hematol. 2005 Dec;84 Suppl 1:61-6. doi: 10.1007/s00277-005-0026-8. PMID 16270213
- [Background] Balbi A, Sottofattori E, Mazzei M, Sannita WG. Study of bioequivalence of magnesium and sodium valproates. J Pharm Biomed Anal. 1991;9(4):317-21. doi: 10.1016/0731-7085(91)80200-s. PMID 1911984
- [Background] Erlich RB, Rickwood D, Coman WB, Saunders NA, Guminski A. Valproic acid as a therapeutic agent for head and neck squamous cell carcinomas. Cancer Chemother Pharmacol. 2009 Feb;63(3):381-9. doi: 10.1007/s00280-008-0747-1. Epub 2008 Apr 9. PMID 18398612
- [Background] Cameron EE, Bachman KE, Myohanen S, Herman JG, Baylin SB. Synergy of demethylation and histone deacetylase inhibition in the re-expression of genes silenced in cancer. Nat Genet. 1999 Jan;21(1):103-7. doi: 10.1038/5047. PMID 9916800
- [Background] Raffoux E, Cras A, Recher C, Boelle PY, de Labarthe A, Turlure P, Marolleau JP, Reman O, Gardin C, Victor M, Maury S, Rousselot P, Malfuson JV, Maarek O, Daniel MT, Fenaux P, Degos L, Chomienne C, Chevret S, Dombret H. Phase 2 clinical trial of 5-azacitidine, valproic acid, and all-trans retinoic acid in patients with high-risk acute myeloid leukemia or myelodysplastic syndrome. Oncotarget. 2010 May;1(1):34-42. doi: 10.18632/oncotarget.106. PMID 21293051
- [Background] Kuendgen A, Bug G, Ottmann OG, Haase D, Schanz J, Hildebrandt B, Nachtkamp K, Neukirchen J, Dienst A, Haas R, Germing U, Gattermann N. Treatment of poor-risk myelodysplastic syndromes and acute myeloid leukemia with a combination of 5-azacytidine and valproic acid. Clin Epigenetics. 2011 Aug;2(2):389-99. doi: 10.1007/s13148-011-0031-9. Epub 2011 Apr 8. PMID 22704349
- [Background] Issa JP, Garcia-Manero G, Huang X, Cortes J, Ravandi F, Jabbour E, Borthakur G, Brandt M, Pierce S, Kantarjian HM. Results of phase 2 randomized study of low-dose decitabine with or without valproic acid in patients with myelodysplastic syndrome and acute myelogenous leukemia. Cancer. 2015 Feb 15;121(4):556-61. doi: 10.1002/cncr.29085. Epub 2014 Oct 21. PMID 25336333
- [Background] Soriano AO, Yang H, Faderl S, Estrov Z, Giles F, Ravandi F, Cortes J, Wierda WG, Ouzounian S, Quezada A, Pierce S, Estey EH, Issa JP, Kantarjian HM, Garcia-Manero G. Safety and clinical activity of the combination of 5-azacytidine, valproic acid, and all-trans retinoic acid in acute myeloid leukemia and myelodysplastic syndrome. Blood. 2007 Oct 1;110(7):2302-8. doi: 10.1182/blood-2007-03-078576. Epub 2007 Jun 27. PMID 17596541
- [Background] Sharma S, Kelly TK, Jones PA. Epigenetics in cancer. Carcinogenesis. 2010 Jan;31(1):27-36. doi: 10.1093/carcin/bgp220. Epub 2009 Sep 13. PMID 19752007
- [Background] Duenas-Gonzalez A, Candelaria M, Perez-Plascencia C, Perez-Cardenas E, de la Cruz-Hernandez E, Herrera LA. Valproic acid as epigenetic cancer drug: preclinical, clinical and transcriptional effects on solid tumors. Cancer Treat Rev. 2008 May;34(3):206-22. doi: 10.1016/j.ctrv.2007.11.003. Epub 2008 Jan 15. PMID 18226465